CLINICAL TRIAL: NCT01690533
Title: Special Drug Use Investigation - Assessment of Efficacy and Safety in Treating Secondary Infection of Chronic Respiratory Disease
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 16515
Record Dates: First submitted 2012-09-19; First posted 2012-09-21 (Estimated); Last update posted 2018-05-21 (Actual); Status verified 2018-05

CONDITIONS: Anti-Infective Agents
Keywords: Avelox; Laryngopharyngitis; Tonsillitis; Bronchitis acute; Pneumonia; Secondary infection in chronic respiratory diseases Sinusitis
MeSH Terms: conditions — Tonsillitis; Bronchitis; Pneumonia | interventions — Moxifloxacin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Avelox (Moxifloxacin, BAY12-8039)

INTERVENTIONS:
Drug: Avelox (Moxifloxacin, BAY12-8039) — Patients treated with Moxifloxacin in daily clinical practice

SUMMARY:
The objective of this study is to assess the efficacy and safety of Avelox Tablet 400 mg (hereinafter as "Avelox") in treating secondary infection of chronic respiratory disease.It is a local prospective and observational study of patients who have received Avelox tablets for Laryngopharyngitis, Tonsillitis, Bronchitis acute, Pneumonia, Secondary infection in chronic respiratory diseases, Sinusitis. A total of 500 patients are to be enrolled and assessed during the period of treatment with Avelox.

ELIGIBILITY:
Inclusion Criteria:

* Patients with secondary infection of chronic respiratory disease (excluding acute bronchitis patients who have been determined to be without chronic respiratory tract disease based on their medical history, x-ray findings, and/or other findings) who meet the following criteria:
* 20 years old or older
* with infection of mild or moderate severity
* Patients who meet the following criteria immediately before starting the therapy: ≥37°C of body temperature, expectoration of purulent or mucopurulent sputum, and either white blood cell count ≥8,000/mm3 or CRP ≥0.7 mg/dL

Exclusion Criteria:

* Patients who are contraindicated based on the product label.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with secondary infection of chronic respiratory disease (excluding acute bronchitis patients who have been determined to be without chronic respiratory tract disease based on their medical history, x-ray findings, and/or other findings)
Sampling Method: Non-Probability Sample
Enrollment: 497 (Actual)
Dates: Start 2008-05-13 (Actual); Primary Completion 2010-12-14 (Actual); Study Completion 2013-07-19 (Actual)

PRIMARY OUTCOMES:
Number of adverse drug reactions (ADRs) and serious adverse events (SAEs) | After 7 days
Clinical efficacy rate (Response, Minor Response, No Response and Indeterminable) assessed by investigator's discretion. Efficacy rate is calculated as number of patients with Response or Minor Response proportional to number of all cases. | After 7 days

SECONDARY OUTCOMES:
ADR incidence rates classified by patient's background factors | After 7 days
Efficacy rates classified by patient's background factors | After 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Multiple Locations, Japan